CLINICAL TRIAL: NCT00104793
Title: Phase II Study of Weekly Irinotecan and Carboplatin in Extensive-Stage Small-Cell Lung Cancer
Brief Title: Irinotecan and Carboplatin in Treating Patients With Newly Diagnosed Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Multinational Trial Organization (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: JMTO-LC02-02; CDR0000415703 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2007-10

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Irinotecan

INTERVENTIONS:
Drug: carboplatin
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving irinotecan together with carboplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving irinotecan together with carboplatin works in treating patients with newly diagnosed extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with newly diagnosed, previously untreated extensive stage small cell lung cancer treated with irinotecan and carboplatin.

Secondary

* Determine the progression-free and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive irinotecan IV and carboplatin IV on days 1 and 8. Treatment repeats every 21 days for 6 courses.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer

  * Extensive stage disease
* Newly diagnosed, treatment-naive disease
* At least 1 unidimensionally measurable lesion
* No massive pleural or pericardial effusion by chest CT scan

  * Manageable effusions allowed

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute granulocyte count ≥ 1,500/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* ALT or AST ≤ 2 times upper limit of normal
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine normal

Cardiovascular

* No myocardial infarction within the past year
* No uncontrolled hypertension
* No unstable angina
* No congestive heart failure
* No ventricular arrhythmia requiring medical intervention
* No other serious cardiovascular disease

Pulmonary

* Arterial oxygen pressure (Pa O_2) ≥ 70 mm Hg
* No interstitial pneumonitis or pulmonary fibrosis by chest x-ray

Other

* Not pregnant or nursing
* No uncontrolled diabetes
* No severe infection
* No paralytic or obstructive ileus
* No serious diarrhea
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix that is in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the chest

  * Other prior radiotherapy allowed

Surgery

* At least 2 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2003-06; Primary Completion 2007-02 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Response

SECONDARY OUTCOMES:
Survival
Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Tadashi Mio, MD, Study Chair — Kyoto University Hospital
Locations (11):
- Japan (11):
  - Gunma Cancer Center, Gunma, Gunma
  - National Hospital Organization - Dohoku National Hospital, Asahikawa, Hokkaido
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - Kurashiki Central Hospital, Kurashiki-shi, Okayama-ken
  - Osaka Kosei Nenkin Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - National Hospital Organization - Osaka National Hospital, Sakai, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Yao Tokusyu-kai General Hospital, Yao, Osaka
  - Tokyo Medical and Dental University, Tokyo, Tokyo
  - National Hospital Organization - Medical Center of Kure, Hiroshima

REFERENCES:
- [Result] Okishio K, Mio T, Kawahara M, Yoshioka H, Yanagihara K, Daimon T, Furuse K. A weekly combination of carboplatin and irinotecan for previously untreated extensive disease small-cell lung cancer, results of a minimum follow-up of 3 years: a multi-center Phase II trial JMTO LC02-02. Jpn J Clin Oncol. 2012 May;42(5):387-93. doi: 10.1093/jjco/hys028. Epub 2012 Mar 19. PMID 22430871